CLINICAL TRIAL: NCT04201457
Title: Phase I/II Trial of Dabrafenib, Trametinib, and Hydroxychloroquine (HCQ) for BRAF V600E-mutant or Trametinib and HCQ for BRAF Fusion/Duplication Positive or NF1-associated Recurrent or Progressive Gliomas in Children and Young Adults
Brief Title: A Trial of Dabrafenib, Trametinib and Hydroxychloroquine for Patients With Recurrent LGG or HGG With a BRAF Aberration
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); American Lebanese Syrian Associated Charities (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-055; UM1CA081457 (NIH); NCI-2019-06216 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-055 (Other: Pediatric Brain Tumor Consortium); PBTC-055 (Other: CTEP)
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Low Grade Glioma (LGG) of Brain With BRAF Aberration; High Grade Glioma (HGG) of the Brain With BRAF Aberration; Low Grade Glioma of Brain With Neurofibromatosis Type 1
Keywords: LGG; HGG; BRAF; NF-1; Autophagy
MeSH Terms: conditions — Glioma | interventions — dabrafenib; trametinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1 Stratum 1 BRAF V600E LGG or HGG (Experimental): LGG or HGG with BRAF V600E/D/K mutation will receive Dabrafenib, Trametinib and Hydroxychloroquine. All medications are administered orally with Dabrafenib and HCQ given twice a day and Trametinib given once per day at the assigned dose for a 28 day course. Courses may repeat until the patient meets an off treatment criteria.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Hydroxychloroquine
- Phase 1 Stratum 2 BRAF aberration or LGG with NF1 (Experimental): LGG with BRAF duplication or fusion with any partner or LGG with NF1 will received Trametinib and Hydroxychloroquine. All medications are administered orally with Trametinib given once per day and HCQ give twice per day at the assigned dose for a 28 day course. Courses may repeat until the patient meets an off treatment criteria.
  Interventions: Drug: Trametinib; Drug: Hydroxychloroquine
- Phase 2 Stratum 3 LGG with BRAF V600 mutation (Experimental): LGG with BRAF V600E/D/K mutation will receive Dabrafenib, Trametinib and Hydroxychloroquine. All medications are administered orally with Dabrafenib and HCQ given twice a day and Trametinib given once per day at the recommended Phase 2 dose for a 28 day course. Courses may repeat until the patient meets an off treatment criteria.
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Hydroxychloroquine
- Phase 2 Stratum 4 HGG with BRAF V600 mutation (Experimental): HGG with BRAF V600E/D/K mutation will receive Dabrafenib, Trametinib and Hydroxychloroquine. All medications are administered orally with Dabrafenib and HCQ given twice a day and Trametinib given once per day at the recommended Phase 2 dose for a 28 day course. Courses may repeat until the patient meets an off treatment criteria
  Interventions: Drug: Dabrafenib; Drug: Trametinib; Drug: Hydroxychloroquine
- Phase 2 Stratum 5 LGG with BRAF aberration (Experimental): LGG with BRAF duplication or fusion with any partner will receive Trametinib and Hydroxychloroquine. All medications are administered orally with Trametinib given once per day and HCQ give twice per day at the recommended Phase 2 dose for a 28 day course. Courses may repeat until the patient meets an off treatment criteria.
  Interventions: Drug: Trametinib; Drug: Hydroxychloroquine
- Phase 2 Stratum 6 LGG with NF Type 1 (Experimental): LGG with Neurofibromatosis Type 1 will receive Trametinib and Hydroxychloroquine. All medications are administered orally with Trametinib given once per day and HCQ give twice per day at the recommended Phase 2 dose for a 28 day course. Courses may repeat until the patient meets an off treatment criteria.
  Interventions: Drug: Trametinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Dabrafenib — Dabrafenib capsule; Dabrafenib Dispersible Tablet
  Other Names: Dabrafenib mesylate; Tafinlar
  Arms: Phase 1 Stratum 1 BRAF V600E LGG or HGG; Phase 2 Stratum 3 LGG with BRAF V600 mutation; Phase 2 Stratum 4 HGG with BRAF V600 mutation
Drug: Trametinib — Tablet; Powder for Oral Solution
  Other Names: Trametinib dimethyl sulfoxide; Mekinist
Drug: Hydroxychloroquine — Tablet
  Other Names: Plaquenil; Plaquinol; Toremonil; Ercoquinn

SUMMARY:
This phase I/II trial is designed to study the side effects, best dose and efficacy of adding hydroxychloroquine to dabrafenib and/or trametinib in children with low grade or high grade brain tumors previously treated with similar drugs that did not respond completely (progressive) or tumors that came back while receiving a similar agent (recurrent). Patients must also have specific genetic mutations including BRAF V600 mutations or BRAF fusion/duplication, with or without neurofibromatosis type 1. Neurofibromatosis type 1 is an inherited genetic condition that causes tumors to grow on nerve tissue. Hydroxychloroquine, works in different ways to stop the growth of tumor cells by killing the cells or stopping them from dividing. Trametinib and dabrafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving hydroxychloroquine with trametinib and/or dabrafenib may lower the chance of brain tumors growing or spreading compared to usual treatments.

DETAILED DESCRIPTION:
In this phase I/II study, the investigators will investigate the safety and efficacy of dabrafenib + trametinib + HCQ (D+T+HCQ) and trametinib + HCQ (T+HCQ) in pediatric and young adult patients with BRAF-altered or NF1-associated gliomas who have previously received a RAF and/or MEK inhibitor. The goal of this study is to optimize the clinical effect of dabrafenib and trametinib by addressing intrinsic and acquired resistance that is well-described in V600E-mutant melanoma and for which there is preclinical and clinical evidence in pediatric gliomas. Aside from overlapping skin toxicity of dabrafenib and trametinib, which preliminarily does not appear worse in the D+T combination in adults and children, potential for ocular toxicity, which has been observed with each agent as monotherapy, will require close monitoring. An important outcome of this study will be improved understanding of resistance mechanisms and the role of autophagy in BRAF-altered or NF1-associated gliomas through sequencing of pre- and post-RAFi or MEKi tumor (when available) and measurement of autophagy inhibition in throughout protocol therapy.

Phase I:

The primary objective of the Phase I component is to estimate the maximum tolerated doses (MTD) and recommended Phase II doses (RP2D) of D+T+HCQ and T+HCQ in children and young adults with recurrent or progressive glioma treated with prior RAF and/or MEK inhibitor therapy.

Patients with BRAF V600E LGG or HGG will receive the combination of D+T+HCQ given orally in the form of capsules which must be taken whole, or an oral solution made from tablets. Hydroxychloroquine will only be administered by oral suspension. Within each combination, Dabrafenib and Hydroxychloroquine will be administered twice a day in a 28-day course. Trametinib will be administered once a day for 28 days during each course. One course is equivalent to 28 days. Therapy with either combination may continue for up to 2 years (26 courses) in the absence of disease progression or unacceptable toxicity.

Phase II Potential patients for the Phase II portion of the trial must provide magnetic resonance imaging studies for central review for screening prior to enrollment: (1) prior targeted MEK/RAF therapy baseline, (2) prior MEK/RAF therapy best response, (3) scan at off treatment, and if different from off treatment (4) scan documenting PD associated with prior MEK/RAF targeted therapy. Additional scans may be requested from the site if the required eligibility assessments cannot be completed based on these minimal imaging requirements.

In the Phase II portion of the trial, patients will continue to receive either the D +T+HCQ or T+HCQ combination at the RP2D defined in the Phase I portion. All drugs will be given continuously without a break unless required for excess toxicity. For Phase I subjects who are treated at the MTD a similar review will take place retrospectively to determine whether the patients meet the criteria to be included in the Phase II cohort.

ELIGIBILITY:
Inclusion Criteria:

* • Patients must have one of the following histologies with molecularly-confirmed diagnosis that is recurrent or progressive. Patients enrolled will be stratified as follows:

  * Phase I:

    * Stratum 1 LGG or HGG with BRAF V600E/D/K mutation
    * Stratum 2 LGG with BRAF duplication or fusion with any partner or LGG with neurofibromatosis type 1
  * Phase II:

    * Stratum 3 LGG with BRAF V600E/D/K mutation
    * Stratum 4 HGG with BRAF V600E/D/K mutation
    * Stratum 5 LGG with BRAF duplication or fusion with any partner
    * Stratum 6 LGG with neurofibromatosis type 1
  * BRAF alterations will be locally determined using molecular methods in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory. Immunohistochemistry for BRAF V600E alone is not adequate and must be confirmed molecularly

    * Phase II patients must have bi-dimensionally measurable disease defined as at least one lesion that can be accurately measured in at least two planes. A target lesion should be chosen
    * Patients are required to have weight >= 9 kg to enroll on any stratum in the Phase I or Phase II
  * Phase I only

    * Patients enrolled on the 8 mg/kg/day (dose level 1) must have a weight < 90 kg
    * Patients enrolled on the 15 mg/kg/day (dose level 2) must have a weight < 80 kg
    * Patients enrolled on the 20 mg/kg/day (dose level 3) must have a weight < 68 kg

      * Patients must have received prior therapy other than surgery and must have fully recovered from the acute treatment related toxicities (defined as =< grade 1) of all prior chemotherapy, immunotherapy, radiotherapy or any other treatment modality prior to entering this study
      * Only applicable to LGG patients on Phase I and all patients on Phase II
  * Patients must have received prior RAF and/or MEK inhibitor therapy and meet one of the following criteria:

    * Did not experience an objective response (defined as < PR) OR
    * Achieved an objective response (CR or PR) but progressed while on active therapy
  * HGG patients on Phase I: may be enrolled regardless of prior MEK /RAF treatment

    • Imaging must be available for central review to confirm eligibility for LGG patients on the Phase I study and all patients on the Phase II study
  * Patients with HGG on the phase I study do not require central imaging review for eligibility
  * Patients with LGG on the Phase I study will not require real-time central imaging review, but imaging must be available for retrospective review in case the subject was enrolled at the RP2D and may be counted as part of the phase II study

    * Patients must have received their last dose of known myelosuppressive anticancer therapy at least 21 days prior to enrollment or at least 42 days if nitrosourea
    * Patient must have recovered from any acute toxicity potentially related to the agent and received their last dose of the investigational or biologic agent >= 7 days prior to study enrollment. For biologic agents or monoclonal antibodies with a prolonged half-life, at least three half-lives must have elapsed prior to enrollment
    * Patients must have had their last fraction of:
  * Craniospinal irradiation, whole brain radiation, total body irradiation or radiation to >= 50% of pelvis or spine >= 6 weeks (42 days) prior to enrollment

    ** Focal irradiation >= 14 days prior to enrollment
    * Patients with neurological deficits should have deficits that are stable for a minimum of 7 days prior to enrollment.
    * Patients with seizure disorders may be enrolled if seizures are controlled. Patients may take non-enzyme inducing anti-epileptic medications
    * Patients who are receiving dexamethasone must be on a stable or decreasing dose for at least 1 week prior to enrollment
    * Karnofsky performance scale (KPS for > 16 years of age) or Lansky performance score (LPS for =< 16 years of age) assessed within 7 days of enrollment must be >= 50
  * Patients who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for assessing the performance score

    * Absolute neutrophil count >= 1.0 x 10^9 cells/ L
    * Platelets >= 100 x 10^9 cells/ L (unsupported, defined as no platelet transfusion within 7 days)
    * Hemoglobin >= 8 g/dl (may receive transfusions)
    * Total bilirubin =< 1.5 times institutional upper limit of normal (ULN)
    * Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 3 x institutional upper limit of normal (ULN)
    * Albumin >= 3 g/dl
    * Serum creatinine based on age/gender. Patients that do not meet these criteria but have a 24-hour creatinine clearance or glomerular filtration rate (GFR) (radioisotope or iothalamate) >= 70 mL/min/1.73 m^2 are eligible
  * Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male); 0.6 (female)
  * Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male); 0.8 (female)
  * Age: 6 to < 10 years; maximum serum creatinine (mg/dL): 1 (male); 1 (female)
  * Age: 10 to < 13 years; maximum serum creatinine (mg/dL): 1.2 (male); 1.2 (female)
  * Age: 13 to < 16 years; maximum serum creatinine (mg/dL): 1.5 (male); 1.4 (female)
  * Age: >= 16 years; maximum serum creatinine (mg/dL): 1.7 (male); 1.4 (female)

    * Left ventricular ejection fraction greater than the institutional lower limit of normal by echo (while not receiving medications for cardiac function)
    * Corrected QT (QTc) =< 480 msec
    * Female patients of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
    * Females of child-bearing potential must use a highly effective method of contraception during dosing of study treatment and for 16 weeks after stopping study medication.
    * Sexually active males must use a condom during intercourse while on study and for 16 weeks after stopping study treatment and agree not to father a child during this period
    * The patient or parent/guardian is able to understand the consent and is willing to sign a written informed consent document according to institutional guidelines

Exclusion Criteria:

* • Breast-feeding women are excluded from this study due to risks of fetal and teratogenic adverse events as seen in animal/human studies

  * Patients with any clinically significant unrelated systemic illness (serious infections or significant cardiac, pulmonary, hepatic or other organ dysfunction), that in the opinion of the investigator would compromise the patient's ability to tolerate protocol therapy, put them at additional risk for toxicity or would interfere with the study procedures or results:

    * Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial. Patients with NF1 and history of plexiform neurofibroma will be permitted to enroll
    * Patients with a previously documented retinal vein occlusion or severe retinopathy
    * Presence of active gastrointestinal (GI) disease or other condition (e.g., small bowel or large bowel resection) that will interfere significantly with the absorption of drugs
  * Patients who are unable to discontinue prohibited medications or herbal preparations within 7 days of enrollment and 14 days of starting study therapy
  * Patients who are receiving any other anti-cancer or investigational drug therapy are ineligible
  * Patients with a history of a known hypersensitivity to dabrafenib, trametinib, HCQ, or any of their excipients or compounds of similar chemical or biologic composition
  * Prisoners will be excluded from this study.
  * Patients who in the opinion of the investigator are unwilling or unable to return for required follow-up visits or obtain follow-up studies required to assess toxicity to therapy or to adhere to drug administration plan, other study procedures, and study restrictions

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD)/ Recommended Phase 2 Dose (RP2D) | Approximately 28 days from start of therapy
  Testing the safety/tolerability of adding HCQ to Dabrafenib + Trametinib or to Trametinib
Maximum Plasma Concentration | 1-4 days
  Maximum plasma concentration Dabrafenib+Trametinib+Hydroxychloroquine or Trametinib +Hydroxychloroquine
Area under the curve (AUC) | 1-4 days
  AUC for Dabrafenib+Trametinib+Hydroxychloroquine or Trametinib +Hydroxychloroquine
Phase II: Sustained objective response rate. | Up to approximately 2 years from the start of therapy
  Number of patients who meet the "better response" criteria, which is a comparison of response on this current protocol therapy versus their best response to previous RAF and/or MEK inhibitor therapy

SECONDARY OUTCOMES:
Phase I: Dose limiting toxicities of D + T HCQ or T + HCQ | course 1 of therapy, approximately 28 days from start of therapy
  Describe the dose limiting toxicities separately for each stratum
Phase I: Response Rate | Up to approximately 2 years from start of therapy
  Proportion of patients who achieve either a partial or a complete response among those with measureable disease at enrollment.
Phase II: Progression-free survival | Start of protocol therapy until progression or last follow-up, up to approximately 2 years from start of treatment
  Time from enrollment up to disease progression or death or loss to follow-up, whichever is first
Phase II: Visual outcome based on Teller Grating Acuity at 55 cm in the left eye in children with tumor involving the visual pathway | Throughout study therapy, up to approximately 2 years from start of therapy
  Teller Grating Acuity at 55 cm in the left eye in children with tumor involving the visual pathway
Phase I and II: Autophagy inhibition as assessed by the accumulation of LC3II in peripheral blood mononuclear cells | Approximately 2 years from start of therapy]
  Accumulation of LC3II in peripheral blood mononuclear cells
Phase I and II: Autophagy inhibition as assessed by the accumulation of p62 in peripheral blood mononuclear cells | Approximately 2 years from start of therapy
  Accumulation of p62 in peripheral blood mononuclear cells
Phase I and II: Presence of MAPK pathway aberrations (other than BRAF) as assessed by whole exome sequencing | At time of study enrollment
  MAPK pathway aberrations (other than BRAF) assessed by whole exome sequencing
Phase I and II: biomarker of resistance to RAF or MEK inhibitor therapy by evaluating matched primary and recurrent/progressive in tumor in plasma (and CSF if clinically indicated) | At enrollment and at the time of every MRI study up to approximately 2 years from the start of therapy
  Evaluating matched primary and recurrent/progressive in tumor in plasma (and CSF if clinically indicated)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Hoffman, DO, Study Chair — Phoenix Children's Hospital
Locations (15):
- United States (15):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - National Cancer Institute Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St. Jude Children Research Hospital, Memphis, Tennessee
  - Texas Children's Cancer Center, Houston, Texas

DOCUMENTS (4):
  • Informed Consent Form: IC Form Phase 1 Stratum 2 (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04201457/ICF_002.pdf
  • Informed Consent Form: IC Form Phase 2 Strata 5 & 6 (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04201457/ICF_004.pdf
  • Informed Consent Form: IC Form Phase 2 Strata 3 & 4 (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04201457/ICF_003.pdf
  • Informed Consent Form: IC Form Phase 1 Stratum 1 (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/57/NCT04201457/ICF_001.pdf